CLINICAL TRIAL: NCT05229601
Title: A Dose Escalation Study of HFB301001 (OX40 Agonist Antibody) in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of HFB301001 in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to discontinue the trial was made as part of a strategic review of the Sponsor's global development portfolio. It is not related to any safety concerns, efficacy findings, recruitment difficulties, or issues with trial conduct.
Sponsor: HiFiBiO Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFB-301001-01; 2021-004854-46 (EudraCT Number)
Record Dates: First submitted 2022-01-19; First posted 2022-02-08 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Soft Tissue Sarcoma; Renal Cell Carcinoma; Uterine Carcinosarcoma; Hepatocellular Carcinoma; Head and Neck Squamous Cell Carcinoma; Melanoma
MeSH Terms: conditions — Sarcoma; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HFB301001 (Experimental): Participants will receive HFB301001 via intravenous infusions
  Interventions: Drug: HFB301001

INTERVENTIONS:
Drug: HFB301001 — Dose Escalation: Participants will be administered dose level 1 in Cohort 1. Participants in Cohorts 2-4 will receive dose levels 2-4, respectively.
  Dose Expansion: Participants with certain cancer types will be administered the dose determined at dose escalation.

SUMMARY:
The purpose of this study is to test the safety and tolerability of HFB301001 in patients with advanced cancers. There are two parts in this study. During the escalation part, groups of participants will receive increasing doses until a safe and tolerable doses of HFB301001 is determined. During the expansion part, participants will take the dose of study drug that was determined from the escalation part of the study and will be assigned to a group based on the type of cancer they have.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, open-label, dose escalation and expansion study in adult patients with advanced cancers. The study will comprise of:

1. A Screening Period of up to 28 days
2. A Treatment Period during which participants will receive the study drug on the first day of each cycle where each cycle is 28 days. Number of cycles depends on how the disease responds to the study drug
3. A Follow-Up Period which involves 1 visit

ELIGIBILITY:
Inclusion Criteria:

* Previously received the following lines of systemic therapy for the advanced/metastatic disease:

  * Soft tissue sarcoma: at least 1 line of therapy
  * Renal cell carcinoma: at least 2 lines of therapy;
  * Uterine carcinosarcoma: at least 1 line of therapy;
  * Hepatocellular carcinoma: at least 1 line of therapy
  * Head and neck squamous cell carcinoma: at least 2 lines of therapy
  * Melanoma:

    * BRAF V600E mutant: must have received at least 2 lines of therapy
    * BRAF V600E wild type: must have received at least 1 line of therapy
* Suitable site to biopsy at pre-treatment and on-treatment
* Measurable disease as determined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-RECIST (iRECIST)
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Exclusion Criteria:

* Systemic anti-cancer therapy within 2 weeks prior to start of study drug.
* For soft tissue sarcoma only: prior immune therapy or immune agonist antibodies
* For uterine carcinosarcoma patients only: prior immune therapy
* Therapeutic radiation therapy within the past 2 weeks
* Prior exposure to agents targeting the OX40 receptor;
* Active autoimmune disease requiring systemic treatment in the previous 2 years;
* Systemic steroid therapy (>10 mg/day of prednisone or equivalent) or any immune suppressive therapy.
* Persisting toxicity of >Grade 1 relating to prior anti cancer therapy with the following exceptions:

  * All grades of alopecia are acceptable;
  * Endocrine dysfunction on replacement therapy is acceptable.
* Severe or unstable medical condition, including uncontrolled diabetes, coagulopathy, or unstable psychiatric condition;
* Major surgery within 2 weeks of the first dose of study drug;
* History or presence of drug or non-drug induced interstitial lung disease or pneumonitis ≥Grade 2;
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to monoclonal antibodies or any excipient of HFB301001;
* Known active malignancy, with the exception of the specific cancer under investigation in this trial, that required treatment within the previous 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious AEs (SAEs), dose-limiting toxicities (DLTs), changes in laboratory values, vital signs and ECG parameters, and tolerability (dose interruptions, reductions, and dose intensity) | Cycle 1 Day 1 to 30 days after the last dose of HFB301001 (each cycle is 28 days)
To determine a Recommended Phase 2 Dose (RP2D) during Dose Expansion | Cycle 1 Day 1 to 30 days after the last dose of HFB301001 (each cycle is 28 days)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST)1.1 and immune-RECIST (iRECIST) | Baseline to 30 days after the last dose of HFB301001 (each cycle is 28 days), assessed up to 3 years
Disease Control Rate (DCR) as determined by RECIST1.1 and iRECIST | Baseline to 30 days after the last dose of HFB301001 (each cycle is 28 days), assessed up to 3 years
Duration of Response (DOR) as determined by RECIST1.1 and iRECIST | Start of first response to first date of disease progression, clinical progression or death, whichever occurs first, assessed up to 3 years
Progression Free Survival (PFS) as determined by RECIST1.1 and iRECIST | Baseline to disease progression or death, whichever occurs first, assessed up to 3 years
Minimum serum concentration (Cmin) | Cycle 1 Day 1 to day of the last dose of HFB301001 (each cycle is 28 days)
Maximum serum concentration (Cmax) | Cycle 1 Day 1 to day of the last dose of HFB301001 (each cycle is 28 days)
Area under the concentration versus time curve (AUC) | Cycle 1 Day 1 to day of the last dose of HFB301001 (each cycle is 28 days)
Terminal half-life (T1/2) | Cycle 1 Day 1 to day of the last dose of HFB301001 (each cycle is 28 days)
Serum concentration for measurement of anti-HFB301001 antibodies | Cycle 1 Day 1 to day of the last dose of HFB301001 (each cycle is 28 days)
To assess the pharmacodynamic (PD) effects of HFB301001 in the blood and in the tumor | Cycle 1 Day 1 to Cycle 3 Day 2 (each cycle is 28 days)
  Percent change in immunologic changes to immune cells in the blood and tumor

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Mayo Clinic, Scottsdale, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NEXT Virginia Cancer Specialists, Fairfax, Virginia
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia